CLINICAL TRIAL: NCT00000107
Title: Body Water Content in Cyanotic Congenital Heart Disease
Status: Completed | Type: Observational
Sponsor: National Center for Research Resources (NCRR) (NIH)
Other Study IDs: NCRR-M01RR00109-0737; M01RR000109 (NIH)
Record Dates: First submitted 2000-01-18; First posted 2000-01-19 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-12

CONDITIONS: Heart Defects, Congenital
Keywords: Cyanotic Congenital Heart Disease
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Case-Control

SUMMARY:
Adults with cyanotic congenital heart disease have elevated levels of plasma proatrial natruretic peptide (proANP) which most likely results in chronic dehydration, leading to reduced oxygen transport to tissues and shortness of breath with activity. The purpose of this study is to characterize adults with cyanotic congenital heart defects with respect to their body composition (water and fat-free mass) and resting metabolic rates. The study consists of several measures of how much body water, fat and lean tissue a subject has, and measures the number of calories the subject's body uses at rest. Adult subjects with cyanotic congenital heart disease will be recruited along with healthy noncyanotic control subjects matched for age, gender, and body weight.

ELIGIBILITY:
Inclusion Criteria:

* Resting blood pressure below 140/90

Ages: 17 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult

CONTACTS AND LOCATIONS:
Locations (1):
- University of Vermont, Burlington, Vermont, United States